CLINICAL TRIAL: NCT00254137
Title: A Randomized Phase II-study to Evaluate the Safety and Efficacy of Capecitabine Plus Irinotecan Plus Cetuximab Compared to Capecitabine Plus Oxaliplatin Plus Cetuximab in First-line Treatment of Patients With Metastatic Colorectal Cancer.
Brief Title: Cap/Iri Plus Cetuximab Compared to Cap/ox Plus Cetuximab in Patients With Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sanofi (Industry); Pfizer (Industry); Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-02-2004
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2004-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: capecitabine; irinotecan; cetuximab; oxaliplatin; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Irinotecan; Oxaliplatin; Cetuximab

INTERVENTIONS:
Drug: capecitabine
Drug: irinotecan
Drug: oxaliplatin
Drug: cetuximab

SUMMARY:
A randomized phase II-study to evaluate the safety and efficacy of capecitabine plus irinotecan plus cetuximab compared to capecitabine plus oxaliplatin plus cetuximab in first-line treatment of patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal cancer.
* EGF-receptor testing.
* No prior chemotherapy for colorectal cancer (except adjuvant chemotherapy with an interval ³ 6 months).
* No prior therapy with topoisomerase-1 inhibitors, no prior therapy directed against the EGF-pathway.
* No prior surgery (except diagnostic biopsy) or radiation therapy 4 weeks before start of study treatment.
* Measurable disease (diameter ³ 20mm, diameter ³ 10mm with spiral-CT).
* Male and female patients ³ 18 years, £ 75 years. Karnofsky PS ³ 70%. Life expectancy ³ 3 months. Effective contraception if risk of conception exists.
* Adequate bone marrow, liver and renal function (leucocytes ³3.000/µl, neutrophils ³1.500/µl, platelets ³100.000/µl, hemoglobin ³9g/dl, bilirubin £1,5x ULN, ASAT and ALAT £3x ULN (£5x ULN with liver metastasis), serum creatinine £1,5x ULN).
* Written informed consent.

Exclusion Criteria:

* Concurrent treatment of colorectal cancer (except study medication).
* EGF-receptor testing not possible.
* Known DPD-deficiency (no particular screening necessary). Known Gilbert-Meulengracht-Syndrome (no particular screening necessary).
* Known or expected contraindication against study medication.
* Participation in other studies during 30 days before study entry.
* Prior myocardial infarction, severe renal insufficiency (creatinine clearance £30ml/min).
* Previous malignancy (except colorectal cancer, history of basal cell carcinoma of skin or pre-invasive carcinoma of the cervix with adequate treatment and no sign of disease during 5 years).
* Known or suspected cerebral metastasis.
* History of inflammatory bowel disease. Symptomatic peritoneal carcinomatosis.
* Drug or alcohol abuse. Lack of adequate legal capacity.
* Breast-feeding or pregnant women.
* Concurrent medication with Sorivudine and analoga, anticoagulation with Cumarine or derivatives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92
Dates: Start 2004-09; Study Completion 2006-11

PRIMARY OUTCOMES:
Objective response rate (CR+PR)

SECONDARY OUTCOMES:
Time to progression.
Disease control rate (CR+PR+SD).
Safety profile.
Grade 3/4- toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, PhD, MD, Principal Investigator — University of Munich - Klinikum Grosshadern